CLINICAL TRIAL: NCT00389298
Title: A Phase 2, Multicenter, Randomized, Double-blinded, and Placebo-controlled Study of the Antiviral Activity, Safety and Pharmacokinetics of VCH-759 in Subjects With Chronic Hepatitis C-infection.
Brief Title: A Proof-of-concept Study of VCH-759 for the Treatment of Hepatitis C-infection.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: ViroChem Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCH759-201
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Viral kinetics; Phase II; Pharmacokinetics (PK); Safety and tolerability
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — VCH-759

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: VCH-759 (BCH-27759)

SUMMARY:
The purpose of this study is to determine whether a 10-day course of therapy with orally administered VCH-759 given at 400-mg, 600-mg or 800-mg three times daily can effectively reduce the amount of circulating virus (i.e., viral load) in patients with early-stage chronic hepatitis C-infection. This study will also evaluate the safety and tolerability of treatment with VCH-759. Blood samples will also be taken to measure the levels of VCH-759 present in plasma at various time points during the treatment period.

DETAILED DESCRIPTION:
The primary objectives of this trial are to assess the antiviral activity, safety, and tolerability of VCH-759 monotherapy in adult subjects with early-stage chronic HCV-infection.

In addition, the pharmacokinetic (PK) profile of VCH-759 at steady state in HCV-infected adults and the relationship between VCH-759 plasma levels and corresponding HCV RNA reduction with the administered dosages of VCH-759 in adults will also be investigated. The kinetics of plasma HCV RNA during treatment for up to ten (10) days with VCH-759 and following discontinuation of therapy will also be studied.

This is a randomized, double-blinded, placebo-controlled study in which subjects will be assigned to receive treatment with one of the following oral dosages of VCH-759: 400 mg t.i.d., 600 mg t.i.d., and 800 mg t.i.d., or placebo; enrollment into the three cohorts will occur sequentially. Within each cohort, subjects will be randomized to a treatment: placebo ratio of 3:1 for a total of 12 subjects per cohort; subjects will be randomized in blocks of 4. The decision to continue dosing within a cohort will be determined by an independent review of all safety data up to and including Day 11 for the first 4 subjects within that dose cohort; this review will be conducted by a qualified medical specialist, in conjunction with the sponsor and medical monitor. The decision to proceed to the next cohort will be decided by an independent review of Day 11 safety data for all 12 subjects in the previous cohort. Eligible subjects will receive study medication three times daily for 10 days and will return to the study center for follow-up assessments on Day 11, Day 17, and Day 24.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age
* Body mass index (BMI) ≤ 30
* No evidence of cirrhosis or have liver fibrosis corresponding to Metavir Stages 0 to 3
* Subject's liver disease is stable (i.e., stable ALT and AST)
* Serologic evidence of chronic hepatitis C-infection (anti-HCV in serum)
* HCV plasma RNA >1 x 105 (copies/mL) at baseline
* HCV Genotype 1
* Documented liver biopsy within the last 5 years
* Hemoglobin > or =11.0 g/dL for females and > or =12.0 g/dL for males
* Platelet count higher than 50
* Treatment-naïve for HCV-infection
* Normal calculated creatinine clearance using the Modification of Diet in Renal Disease (MDRD) study formula
* Normal thyroid function
* Female subjects, cannot be pregnant or breastfeeding and must be either postmenopausal, surgically sterile, abstinent, or using two proven methods of birth control
* Sexually active male subjects, must be practicing acceptable methods of contraception (vasectomy, use of condom plus spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period
* Negative serum ß-HCG (females only)
* Provided informed consent
* Willing to comply with all study requirements

Exclusion Criteria:

* Participating in any other clinical studies or have participated in another clinical trial within the last 30 days
* Have relapsed following previous therapy for hepatitis C-infection
* Actively taking hard illicit drugs (such as cocaine, phencyclidine, or crack within 6 months before screening visit)
* Evidence of liver cirrhosis
* Child-Pugh score >5
* Any cause of liver disease other than chronic hepatitis C-infection, including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Autoimmune thyroidopathy
  * Alcoholic liver disease
  * Nonalcoholic steatohepatitis
  * Drug-related liver disease
  * Active malignant disease or suspicion or history of malignant disease within five previous years (except for adequately treated basal cell carcinoma)
* Organ transplants, except for corneal or hair transplant
* Clinically significant electrocardiogram abnormalities and/or cardiovascular dysfunction within 6 previous months (e.g., angina, congestive heart failure, recent myocardial infarction, significant arrhythmia, or prolongation of QTc interval)
* Significant renal, pulmonary, gastrointestinal absorption, or neurological diseases, or neoplasia
* Type 1 diabetes, or Type II diabetes being treated with oral hypoglycemic agents
* Co-infection with hepatitis B (HBV) and/or human immunodeficiency (HIV) virus
* Taking the following concomitant medications:

  * Drugs of abuse (as outlined above)
  * Systemic antibiotic, antiviral, or antifungal treatments
  * All cytostatic or oncolytic medications
  * Drugs that are under routine therapeutic drug monitoring such as antiepileptic (anti-seizure) drugs, digoxin, coumadin and others
  * All lipid lowering agents
  * Drugs that influence hemostasis
  * Thyreostatic drugs from the group of thionamids
  * The following antihistaminics: terfenadine, cyproheptadine and promethazine
  * Tricyclic antidepressants
  * Antipsychotic drugs (neuroleptics)
  * Lithium
  * Thalidomide
* Other condition that, in the investigator's opinion, could determine that the subject's participation in the study is not indicated or could interfere with the subject's participation in and completion of study
* Randomized to this study more than once

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in baseline HCV plasma RNA (i.e., viral load) at Day 11.

SECONDARY OUTCOMES:
The change in plasma HCV RNA (i.e., viral load) over the treatment period (Days 1 to 10 will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Petrella, M.Sc., Ph.D., Study Director — ViroChem Pharma
Locations (4):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - Ottawa Hospital; General Campus, Ottawa, Ontario
  - McGill University Hospital Centre (MUHC) - Royal Victoria Hospital, Montreal, Quebec